CLINICAL TRIAL: NCT06874712
Title: Interest of LC-OCT for Diagnosing Inflammatory Dermatoses: Comparison of Images Obtained with LC-OCT and Those from Histological Sections "ODIN (OCT Dermatoses INflamaatoires)
Brief Title: Interest of LC-OCT for Diagnosing Inflammatory Dermatoses: ODIN (OCT Dermotoses INflammatoires)
Acronym: ODIN
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5184
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Skin Disease, Psoriasiform Dermatoses, Eczematiform Dermatoses, Lichenoid Dermatoses, Psoriasis, Eczema, Lichen, Lupus, Dermatomyositis
MeSH Terms: conditions — Dermatitis; Psoriasis; Eczema; Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (3):
- Definitive histopathological diagnosis of eczematiform dermatosis
- Psoriasiform dermatosis
- Lichenoid dermatosis

SUMMARY:
Inflammatory dermatoses (eczematiform dermatoses, psoriasiform dermatoses, lichenoid dermatoses, toxic dermatoses, auto-immune and auto-inflammatory dermatoses, etc.) and their differential diagnoses (infectious or para-infectious dermatoses, deficiency dermatoses, etc.) are frequent reasons for dermatology consultations. These dermatoses are clinically heterogeneous eruptions for which a skin biopsy for histological examination may be routinely required to confirm the diagnosis.

LC-OCT (DeepLive Damae Medical machine) is a new non-invasive skin imaging technique (using non-ionizing infrared light), enabling observation of skin tissue to a depth of 500 µm with a resolution of 1 µm (= "cellular" resolution, the keratinocyte, the main skin cell, measuring between 5 and 10 µm).

This technique has already proved its worth in the diagnosis of skin cancers, and has the advantage of being non-invasive, painless and quicker than a biopsy. The investigators of the study want to study its value in the diagnosis of inflammatory dermatoses.

During the consultation dedicated to skin biopsy, a cutaneous LC-OCT examination is routinely performed, but only for exploratory purposes, allowing better targeting of the most modified area. The aim of the study is to describe and analyze the characteristics of cutaneous imaging (LC-OCT) in inflammatory dermatoses, comparing them with the histological appearance of biopsy specimens.

This is a preliminary study aimed at defining the value of LC-OCT in the diagnosis of inflammatory dermatoses, in the hope of replacing skin biopsy in the future.

ELIGIBILITY:
Inclusion Criteria:

* - Age greater than or equal to 18 years.
* Definitive histopathological diagnosis of inflammatory dermatosis, including classification by type (eczematiform, psoriasiform or lichenoid) and subtype (e.g. atopic dermatitis for eczematiform dermatosis, lupus for lichenoid dermatosis, etc.).
* Availability of good-quality LC-OCT images/videos, with at least one interpretable 3D block, a video scanning lesional and healthy skin in a manner deemed "sufficient", as judged collegially by the authors.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a definitive histopathological diagnosis of inflammatory dermatosis with a classification by type (eczematiform, psoriasiform or lichenoid)
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Describe presence or absence of signs of inflammatory dermatoses found on LC-OCT images and on histological sections, in the same patient. | Baseline (day of realisation of the two examinations).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Dermatologie, HEH, HCL, France, France